CLINICAL TRIAL: NCT02542150
Title: Effects of Acetate and Alcohol on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 15-0933; UL1TR001082 (NIH)
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Blood Flow; Brain Function
MeSH Terms: interventions — Acetates; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- acetate arm (Experimental): IV acetate given during magnetic resonance scan
  Interventions: Drug: acetate
- alcohol arm (Experimental): jello shots given before magnetic resonance scan
  Interventions: Drug: alcohol

INTERVENTIONS:
Drug: acetate — acetate infusion, saline infusion, functional magnetic resonance imaging (fMRI) scan
  Other Names: ethanoate
  Arms: acetate arm
Drug: alcohol — a "jello shot" containing alcohol, a jello shot containing no alcohol, fMRI scan.
  Other Names: ethanol
  Arms: alcohol arm

SUMMARY:
This study plans to learn more about how alcohol and its metabolite, acetate, affect the brain.

DETAILED DESCRIPTION:
This study plans to learn more about how alcohol and its metabolite, acetate, affect brain function.

ELIGIBILITY:
Inclusion Criteria-all:

1. Subjects who are age 21-55,
2. Subjects who are proficient in English ,
3. Subjects who understand the nature of the study,
4. Subjects who have signed an informed consent,
5. Subjects who are non-smoking (defined as fewer than 20 cigarettes lifetime),

Inclusion Criteria-moderate drinkers:

1. Subjects who are moderate drinkers (male:1-14 drinks per week; female: 1-7 drinks per week).
2. Subjects who have drunk at least 2 drinks in one hour in the past, and have no history of dependence on drugs or alcohol

Inclusions-AUD:

(1) Subjects who meet DSM-V criteria for lifetime history of Alcohol Use Disorder (AUD)

Exclusion Criteria-all:

1. Subjects who have a "facial flushing" response to alcohol,
2. Subjects who are pregnant or nursing,
3. Subjects who have major medical problems including diabetes, high blood pressure (> 150/90), prior neurological or psychiatric history (schizophrenia, bipolar, or current major depressive disorder), epilepsy (alcohol withdrawal seizures is not an exclusion),
4. Subjects who have been told they have or been diagnosed with liver or kidney disease,
5. Subjects who have chronic gastrointestinal disease,
6. Subjects who are obese (BMI>30 kg/m2),
7. Subjects who take psychoactive medications,
8. Subjects who have prior head trauma resulting in loss of consciousness >15 minutes,
9. Subjects who have Magnetic Resonance (MR) exclusions which include claustrophobia, intracranial, orbital, or spinal metal implants, pacemakers, cochlear implants, cardiac stents or other non-MR-compatible implants or devices.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody L Tanabe, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tanabe J, Yamamoto DJ, Sutton B, Brown MS, Hoffman PL, Burnham EL, Glueck DH, Tabakoff B. Effects of Alcohol and Acetate on Cerebral Blood Flow: A Pilot Study. Alcohol Clin Exp Res. 2019 Oct;43(10):2070-2078. doi: 10.1111/acer.14173. Epub 2019 Aug 24. PMID 31386214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates: January 2016-March 2017 Target population: Healthy controls Method: Advertisements, flyers, word of mouth
Groups:
- Acetate Arm: Placebo for 1 hour, then Acetate for 1 hour
  IV acetate given during magnetic resonance scan.
  acetate: acetate infusion, saline infusion, functional magnetic resonance imaging (fMRI) scan
- Alcohol Arm: Placebo for 1 hour, then Alcohol (given as a single dose of jello).
  jello given before magnetic resonance scan
  alcohol: jello containing alcohol, jello containing no alcohol, fMRI scan.
Period: Overall Study
Arm/Group | Acetate Arm | Alcohol Arm
Started | 12 | 12
Completed Placebo | 12 | 12
Started Intervention | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acetate Arm: Placebo for 1 hour, then Acetate for 1 hour.
  IV acetate given during magnetic resonance scan
  acetate: acetate infusion, saline infusion, functional magnetic resonance imaging (fMRI) scan
- Alcohol Arm: Placebo for 1 hour, then alcohol (given as a single dose with jello).
  jello given before magnetic resonance scan
  alcohol: jello containing alcohol, jello containing no alcohol, fMRI scan.
- Total: Total of all reporting groups
Arm/Group | Acetate Arm | Alcohol Arm | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.2) | 31.1 (3.9) | 28.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebral Blood Flow as Measured With Arterial Spin Labeling
Description: cerebral blood flow is measured during a functional magnetic resonance imaging (fMRI). The reported data reflects best efforts to quantify the collected image data.
Time Frame: fMRI scan will be scheduled for 1-3 weeks after enrollment. Total visit will be about 6 hrs.
Measure: Mean (Standard Deviation); unit: cc/100 mg/min
Groups:
- IV Placebo (Acetate Arm): Placebo given before Acetate.
- Oral Placebo (Alcohol Arm): Placebo given before Alcohol.
Arm/Group | Acetate Arm | IV Placebo (Acetate Arm) | Alcohol Arm | Oral Placebo (Alcohol Arm)
Number analyzed (Participants) | 12 | 12 | 12 | 12
cc/100 mg/min
  Right Thalamus | 31.7 (5.6) | 26.9 (5.7) | 30.0 (9.7) | 25.0 (7.5)
  Left Thalamus | 32.8 (6.8) | 27.3 (5.6) | 29.9 (8.9) | 24.9 (6.7)

ADVERSE EVENTS:
Time Frame: 1 Day
Groups:
- Alcohol Arm: jello given before magnetic resonance scan
  alcohol: jello containing alcohol, jello containing no alcohol, fMRI scan.
Arm/Group | Acetate Arm | IV Placebo (Acetate Arm) | Alcohol Arm | Oral Placebo (Alcohol Arm)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12 | 0/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetate Arm (N=12) | IV Placebo (Acetate Arm) (N=12) | Alcohol Arm (N=12) | Oral Placebo (Alcohol Arm) (N=12)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data collection for an outcome measure related to brain activity during decision making before and after receiving alcohol or acetate was never completed due to feasibility and funding limitations and challenges encountered during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02542150/Prot_SAP_000.pdf